CLINICAL TRIAL: NCT01545674
Title: Prenatal Non-invasive Aneuploidy Test Utilizing SNPs Trial (PreNATUS)
Brief Title: Prenatal Non-invasive Aneuploidy Test Utilizing SNPs Trial
Acronym: PreNATUS
Status: Terminated | Type: Observational
Why Stopped: Non-invasive Prenatal Screening CLIA test performance validated in other cohort. Decided samples not required, study aims achieved through other studies.
Sponsor: Natera, Inc. (Industry)
Collaborators: Columbia University (Other); George Washington University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: GSN012B; 1R44HD062114 (NIH)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Trisomy 13; Trisomy 18; Trisomy 21; Aneuploidy
Keywords: Aneuploidy; Non-invasive Prenatal Diagnosis; Prenatal Blood Test; Prenatal Aneuploidy Screening; Trisomy 13; Trisomy 18; Trisomy 21; Trisomy; Down Syndrome; Turner Syndrome; Edwards Syndrome
MeSH Terms: conditions — Trisomy 13 Syndrome; Trisomy 18 Syndrome; Down Syndrome; Aneuploidy; Trisomy; Turner Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Sample Prepared DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnant Women Blood Draw: Pregnant Women with elevated risk of trisomic pregnancy to donate a blood sample through one time blood draw
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Blood will be drawn from the mother and father

SUMMARY:
This prospective blinded study will assess the diagnostic capability of an informatics enhanced SNP based technology (Parental Support) to identify pregnant women who are carrying a fetus with an aneuploidy from fee floating DNA in the maternal blood.

DETAILED DESCRIPTION:
First trimester screening is the current standard of care for pregnant women in the United States. Women with a high screening risk for trisomy then have invasive testing, which carries a risk of miscarriage, to definitively determine if the fetus has trisomy. Because of the high false negative rate of the first trimester screening, an unacceptable number of trisomic fetuses are not detected. Moreover, because of the high false positive rate, an unacceptable number of women undergo invasive follow up testing. Additional screening tests are needed that combine a high sensitivity, a low false positive rate, and minimal or no risk to the fetus.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy
2. Gestational age between 8 weeks 0 days and 23 weeks, 6 days by best obstetrical estimate
3. Mother has a high or moderate risk for trisomy
4. Mother is planning to have or has had an amniocentesis or chorionic villus sampling (CVS) procedure

Exclusion Criteria:

1. Unavailability of the father to provide a genetic sample (e.g. sperm donor, non-paternity)
2. Egg donor used
3. Mother or father have known chromosomal abnormalities (including known balanced translocations)
4. Participation in the study in a previous pregnancy
5. Pregnancy is a result of IVF with pre-implantation genetic diagnosis

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant Women
Sampling Method: Non-Probability Sample
Enrollment: 937 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the test to diagnose aneuploidy in a fetus at chromosomes 13, 18, 21, X and Y. | Between first trimester screening (10-14 weeks GA) and invasive testing (amniocentesis or CVS).
  The primary objective is to determine the diagnostic capability of the test to detect autosomal aneuploidy (chromosomes 13, 18, 21) and sex aneuploidy (X and Y).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wapner, MD, Principal Investigator — Columbia University
Locations (29):
- United States (24):
  - University of Alabama, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Adventist Hinsdale Hospital, Hinsdale, Illinois
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - NY Methodist Hospital, Brooklyn, New York
  - Madonna Perinatal, Mineola, New York
  - New York University, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Columbia University, New York, New York
  - Carnegie Imaging for Women, New York, New York
  - Montefiore Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Mt Sinai Hospital, Toronto, Canada
- Royal College of Surgeons in Ireland, Dublin, Ireland
- University of Perugia, Perugia, Italy
- Hamchoon Women's Clinic, Seoul, South Korea
- Institut Universitari Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
A peer reviewed publication is planned from this study.